CLINICAL TRIAL: NCT02477345
Title: Compassionate Use of Omegaven IV Fat Emulsion
Status: No longer available | Type: Expanded Access
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jonathan Blau, PI, Northwell Health
Other Study IDs: SIUH12-025
Record Dates: First submitted 2013-11-27; First posted 2015-06-22 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Cholestasis; Liver Disease
Keywords: Cholestasis; Parenteral Nutrition; Liver disease
MeSH Terms: conditions — Cholestasis; Liver Diseases; Hyperphagia | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Omegaven IV — Omegaven will be initiated at a dose of 0.5 gram/Kg/day and is infused over 24 hours for 1-2 days, and then advanced to
  1 gram/Kg/day. Omegaven will be infused intravenously through either a central or peripheral catheter alone or in conjunction with parenteral nutrition. Omegaven will continue until weaned from PN. Monotherapy with Omegaven can continue as an additional source of calories after the dextrose/protein portion of PN is discontinued. Omegaven may be restarted within seven days of discontinuing therapy. After seven days, and meeting inclusion criteria, Omegaven can resume at the initial dose of 0.5 grams/Kg/day, advancing to 1 gm/kg/day.
  Other Names: Fat Emulsion

SUMMARY:
This protocol involves the compassionate use of intravenous fish oil infusion, Omegaven. The protocol involves infants and children with parenteral nutrition-associated liver disease to enable the reversal of elevated serum liver enzymes and direct bilirubin (cholestasis).

DETAILED DESCRIPTION:
In the United States, patients dependent upon parenteral nutrition (PN) receive parenteral fat emulsions composed of soybean oils. Lipids are necessary in PN dependent patients due to their high caloric value and essential fatty acid content. Intravenous lipid emulsions have been implicated in predisposing patients to PN associated liver disease. Phytosterols such as those contained in soybean oils are thought to have a deleterious effect on biliary secretion. Accumulation of lipids in the hepatic Kupffer cells may further impair liver function.

Omega 6 fatty acid emulsions prevent fatty acid emulsions prevent fatty acid deficiency, it is thought that they are not cleared in a manner similar to enteral chylomicrons and therefore accumulate in the liver and resulting in steatotic liver injury (neonatal cholestasis). It is hypothesized that a fat emulsion comprised of omega 3 fatty acids (i.e.: fish oil), such as de novo lipogenesis, the reduction of arachidonic acid-derived inflammatory mediators, prevention of essential fatty acid deficiency through the presence of small amounts of arachidonic acid, and improved clearance of lipids from the serum. Animal studies have shown that IV fat emulsions such as fish oil that are high in eicosapentaenic and docosahexaenoic acid reduce impairment of bile flow which is seen in cholestasis caused by conventional fat emulsions. Furthermore, intravenous omega-e fatty acids are well tolerated and might reduce the hepatic dysfunction. By administering Omegaven in place of conventional phytosterol/soybean fat emulsion, the progression of PN-associated cholestasis can be prevented or reversed.

ELIGIBILITY:
Inclusion Criteria:

* subjects will be infants and children from birth to 5 years of age
* diagnosis of parenteral nutrition associated liver disease (PNALD) (defined as two consecutive direct bilirubin levels of 2 mg/dl or more) in a parenteral nutrition-dependent infant or child.
* subject must have utilized standard therapies to prevent the progression of the cholestasis including reduction/removal of copper and manganese from daily PN, trial of enteral feedings if possible, and the use of ursodiol and/or phenobarbital.

Exclusion Criteria:

* patients are excluded if they have other documented causes of chronic liver disease (i.e.: Hepatitis C, cystic fibrosis, biliary atresia, alpha-1-anti-trypsin deficiency),
* or already have signs of proven severe advanced liver disease including cirrhosis on biopsy, varices, ascites.

Additional exclusion criteria:

* an active coagulopathy characterized by ongoing bleeding or by a requirement for clotting factor replacement (e.g. fresh frozen plasma or cryoprecipitate) to maintain homeostasis
* impaired lipid metabolism
* severe hyperlipidemia with or without pancreatitis
* unstable diabetes mellitus
* hyperglycemia
* stroke, embolism
* collapse and shock
* recent myocardial infarction (MI)
* cholestasis due to any reason other than parenteral nutrition associated cholestasis (PNAC)
* active new infection at time of initiation of Omegaven
* hemodynamic instability
* patient cannot be enrolled in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Blau, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

DOCUMENTS (3):
  • Study Protocol (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT02477345/Prot_000.pdf
  • Informed Consent Form (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT02477345/ICF_001.pdf
  • Statistical Analysis Plan (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT02477345/SAP_002.pdf